CLINICAL TRIAL: NCT03293940
Title: Percutaneous Image Guided Cryoablation of the Intercostobrachial Nerve for Management of Post Mastectomy Pain Syndrome
Brief Title: Cryoablation for Post Mastectomy Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, John Prologo, Assistant Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00094527
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Post-Mastectomy Chronic Pain Syndrome (Disorder)
Keywords: Breast Pain; Nerve Pain; Mastectomy; Lumpectomy; Breast Reconstruction
MeSH Terms: conditions — Mastodynia; Neuralgia | interventions — Cryosurgery; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoablation Group (Experimental): After an initial diagnostic visit to locate the pain causing nerve, participants randomized to this arm will receive the cryoablation procedure.
  Participants will have the option to crossover to tPNB 90 days post the initial intervention.
  Interventions: Procedure: Cryoablation
- Control Group (Active Comparator): After an initial diagnostic visit to locate the pain causing nerve, participants randomized to this arm will receive the nerve block procedure.
  Participants will have the option to crossover to cryoablation treatment 90 days post the initial intervention.
  Interventions: Procedure: Therapeutic Peripheral Nerve Block (tPNB) Injection

INTERVENTIONS:
Procedure: Cryoablation — The cryoablation procedure, a needle will be inserted and directed toward the target pain area. More than one needle may need to be used. A CT scan will be done during the procedure to help guide the needle which will be held in position by the study doctor(s) once it reaches the target area. With the needle(s) in place, the study doctor(s) will freeze the nerve over 5 minutes. A 3 minutes thaw will follow, then a second 5 minutes freeze and a final 3minute thaw. This portion of the procedure can last from 25 to 45 minutes. Once the nerve has been properly treated, the cryoablation needle(s) will be withdrawn.
  Arms: Cryoablation Group
Procedure: Therapeutic Peripheral Nerve Block (tPNB) Injection — During the nerve block procedure, a needle will be inserted and directed toward the target pain area. More than one needle may need to be used. A CT scan will be done during the procedure to help guide the needle which will be held in position by the study doctor(s) once it reaches the target area and anesthetic will be injected into the targeted area.
  The tPNB injection consists of 4 cc of 0.25% Bupivicaine and 1 cc of 6mg/ml betamethasone.
  Arms: Control Group

SUMMARY:
This is a prospective, randomized, parallel-group, treatment control trial with cross-over options performed at four sites. The purpose of this study is to assess the efficacy and safety of cryoablation therapy for the treatment of post mastectomy pain syndrome.

DETAILED DESCRIPTION:
This is a prospective, randomized, parallel-group, treatment control trial with cross-over options performed at four sites. The purpose of this study is to assess the efficacy and safety of cryoablation therapy for the treatment of post mastectomy pain syndrome.

Participants will be randomized to receive cryoablation or a therapeutic peripheral nerve block injection (tPNB). All participants will be evaluated at baseline and after treatment at 10 days, 90 days, and 180 days via clinical visits.

The option to undergo cryoablation or tPNB will be offered to all participants at the end of the 90 day post-procedure assessment. Each subject that elects the crossover intervention will be assessed over the same time period and in an identical fashion to the initial intervention, including a final long term follow up (LTFU) assessment at 180 days post-cryoablation.

ELIGIBILITY:
Inclusion Criteria:

* Status post breast surgical intervention, to include mastectomy, partial mastectomy, lumpectomy, or reconstruction
* Persistent pain in the distribution of the Intercostobrachial nerve: the residual breast, surgical bed, ipsilateral medial arm, and/or axilla following tissue healing (> 1 month postoperative)
* Positive response to local anesthetic nerve block, performed under imaging guidance. A positive response is defined as a ≥ 3 point change on a standard 11 point visual analog scale (VAS)
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Active infection
* Underlying cervical segmentation or other cervical spinal anomaly that results in differential nerve root pressures
* Immunosuppression
* Uncorrectable coagulopathy
* Currently pregnant, nursing or planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Change in Breast Pain Intensity assessed by the Visual Analog Scale (VAS) Score | Baseline, Post-Intervention (24 Hours)
  Participants' ratings of perceived pain intensity will be captured with the VAS, a 10cm horizontal line with the extremes labeled, "No pain" and "Worst Possible Pain. Participants mark a point along the continuum and it is scored by measuring the distance, in mm, from the "no pain" end to the participant's mark. A greater the distance from the "no pain" mark to the participants mark indicates greater pain.
Change in Numerical Rating Scale (NRS) of Pain Intensity Score | Baseline, Post-Intervention (24 Hours)
  The NRS is an 11-point rating scale with 0 = "No Pain" and 10 = "Pain as bad as you can imagine". Total scores range from 0-10 points, with higher scores indicating greater pain intensity.

SECONDARY OUTCOMES:
Patient Global Impression of Change Scale (PGIC) Score | Post-Intervention (Up to 24 Hours)
  The PGIC is a comprehensive, single-item estimate of treatment-related improvement that asks participants to consider their current status compared to pre-treatment and rate it on a 7-point scale (very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse). Total scores range from 1 to 7; 1 representing no change and 7 representing considerable improvement.
Brief Pain Inventory Short Form (BPI) Score | Post-Intervention (Up to 24 Hours)
  The BPI captures two broad pain domains: 1) the sensory intensity of pain, and 2) the degree to which pain interferes with different areas of life. Scores are based on the two domains: the pain severity score is the mean of items 3-6 (pain at its worst, pain at its least). The pain interference score is the mean of items 9A-9G (interference of pain with: general activity, mood, walking, normal work, relations, sleep,enjoyment of life). Higher pain scores indicate greater pain and greater interference with daily activities.
McGill Pain Questionnaire Short Form 2 (MPQ) Score | Post-Intervention (Up to 24 Hours)
  The MPQ consists of 24 assessments: 22 questions list a qualitative description of pain symptoms that patients may have felt during the past week and 1 question evaluates present pain intensity, both of which are rated on a numerical rating scale with 0= "None" and 10= "Worst Possible"; the final question evaluates the patient's overall total pain experience on a 6-item scale (no pain, mild, discomforting, distressing, horrible, excruciating). Total scores are on a continuum. The higher the total score, the pain experience for the participant increases.

OTHER OUTCOMES:
Lost to Follow Up Rate | Duration of Study (Up to 180 Days)
  The number of participants who cannot be contacted prior to completing all study visits.
Death Rate | Duration of Study (Up to 180 Days)
  The number of deaths that occur throughout the duration of the study.
Participant Withdrawal Rate | Duration of Study (Up to 180 Days)
  The number of participants who withdraw from the study prior to completing all visits and after providing consent for participation.
Declination Rate | Duration of Study (Up to 180 Days)
  The number of eligible participants who decline study participation after being approached to participate.
Screen Failure Rate | Duration of Study (Up to 180 Days)
  The number of participants who are not eligible for study participation after conducting screening procedures.
Percent Post Mastectomy Participants Enrolled | Post Study Completion (Up to 2 Years)
  Of the total number of post mastectomy patients at all sites, the percentage of patients who have consented to study participation.
Participant Retention Rate | Duration of Study (Up to 180 Days)
  The number of participants who sign consent and complete all study visits.
Total Recruitment Number | Duration of Study (Up to 180 Days)
  The total number of participants recruited to the study.
Frequency of Breakthrough Pain Events | Duration of Study (Up to 180 Days)
  The frequency of breakthrough pain events that require emergency or rescue analgesic use measured in hours.
Number of Breakthrough Pain Events | Duration of Study (Up to 180 Days)
  The number of breakthrough pain events that require emergency or rescue analgesic use reported during study visits.
Proportion of Participants that Experience Adverse Events | Duration of Study (Up to 180 Days)
  The number of participants who experience adverse events divided by the total number of participants.

CONTACTS AND LOCATIONS:
Overall Officials: John Prologo, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Emory St. Joseph's Hospital, Atlanta, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia